CLINICAL TRIAL: NCT01229150
Title: Randomized Phase II Study of AZD6244 MEK-Inhibitor With Erlotinib in KRAS Wild Type and KRAS Mutant Advanced Non-Small Cell Lung Cancer
Brief Title: Randomized Phase II Study of AZD6244 (Mitogen-activated Protein Kinase Inhibitor) MEK-Inhibitor With Erlotinib in KRAS Wild Type Advanced Non-Small Cell Lung Cancer (NSCLC) and a Randomized Phase II Study of AZD6244 With Erlotinib in Mutant KRAS Adva...
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: University of California, Davis (Other); University of Chicago (Other); University of Southern California (Other); City of Hope Medical Center (Other)
Responsible Party: Principal Investigator, Arun Rajan, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100218; 10-C-0218; NCT01239290 (obsolete NCT alias)
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Non Small Cell Lung Carcinoma
Keywords: Kinase Signal Transduction Pathway; Tumor Mutational Analysis; Tissue Immunohistochemistry; MIB-1 (Ki-67) Rate; PERK Level; Lung Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — AZD 6244; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- KRAS Mut 2 (Active Comparator): KRAS Mutant patients randomized to combination therapy arm
  Interventions: Drug: AZD6244 + Erlotinib
- KRAS Mut 1 (Active Comparator): KRAS Mutant patients randomized to monotherapy arm
  Interventions: Drug: AZD6244
- WT KRAS 1 (Active Comparator): Wild-Type KRAS patients randomized to monotherapy arm
  Interventions: Drug: Erlotinib
- WT KRAS 2 (Active Comparator): Wild-Type KRAS patients randomized to combination therapy arm
  Interventions: Drug: AZD6244 + Erlotinib

INTERVENTIONS:
Drug: AZD6244 — For KRAS mutant patients randomized to the single agent arm, AZD6244 75 mg bid (twice a day).
  Arms: KRAS Mut 1
Drug: Erlotinib — For Wild-Type KRAS patients randomized to the single agent arm, Erlotinib 150 mg qd (every day)
  Arms: WT KRAS 1
Drug: AZD6244 + Erlotinib — For KRAS mutant patients and Wild-Type KRAS patients randomized to the combination arm (arms are stratified based on KRAS mutational status), AZD6244 150 mg qd (every day) + erl (erlotinib) mg qd.
  Arms: KRAS Mut 2; WT KRAS 2

SUMMARY:
Background:

AZD6244 (ARRY-142886) is an investigational anticancer drug that is designed to block a critical component (MEK (methyl ethyl ketone)) of a pathway (MAP (mitogen-activated protein) kinase pathway) that causes some lung cancer cells to grow. The MAP kinase pathway could be overactive in a proportion of lung cancers, including some which also have another mutation in a protein known as KRAS (Kirsten rat sarcoma viral oncogene homolog). Approximately 20% of lung cancers have KRAS mutations which can make some cancer treatments including erlotinib, a standard anticancer treatment drug less effective. Researchers are interested in determining whether AZD6244 is effective in treating advanced NSCLC (non small cell lung cancer), including KRAS mutated lung cancer that has not responded to standard therapy.

Objectives:

To determine the effectiveness of AZD6244, either alone or in combination with erlotinib, in preventing tumor growth in individuals with NSCLC.

Eligibility:

Individuals at least 18 years of age who have been diagnosed with advanced NSCLC that has not responded to standard therapy.

Design:

* Participants will be screened with a medical history, physical examination, blood tests, imaging studies, and potentially, tumor biopsy tests to determine whether a participant's NSCLC contains mutations in the KRAS protein.
* Participants will be divided into two groups based on the status of the KRAS protein in their NSCLC tumor cells:
* Individuals with normal KRAS protein: Half will receive AZD6244 and erlotinib, and half will receive only erlotinib.
* Individuals with mutated KRAS protein: Half will receive AZD6244 and erlotinib, and half will receive only AZD6244.
* Participants will take their assigned medications daily (on an empty stomach in the morning and/or evening, depending on the treatment) for 28-day cycles of treatment. Participants will also keep a medication diary to record any side effects.
* Participants will have frequent blood tests during the first cycle of treatment, and will have imaging studies or other tests as required by the study researchers. Participants may also have an additional tumor biopsy after the end of the first treatment cycle.
* Treatment will continue until the disease progresses, significant side effects develop, the participant chooses to leave the study, or the researchers end the study....

DETAILED DESCRIPTION:
Background:

Lung Cancer is the leading cause of death among both men and women. Of the approximately 172,000 patients that are diagnosed every year with non small cell lung cancer (NSCLC) in the US, 55% present with advanced stage disease. The current treatment for advanced NSCLC is first line chemotherapy with a platinum-based doublet. Second line treatment for recurrent or progressive disease includes treatment with chemotherapy or treatment with an oral EGFR (epidermal growth factor receptor) tyrosine kinase inhibitor. Several mechanisms of resistance to EGFR tyrosine kinase inhibitors have been discovered. Presence of KRAS mutations is one of them. AZD6244 (ARRY-142886) is an investigational drug that is orally available and targets the critical kinase (MEK) in the mitogen-activated protein (MAP) kinase signal transduction pathway which is activated in NSCLC and is downstream of EGFR.

Objectives:

* Determine the progression free survival (PFS) using the combination of AZD6244 and erlotinib in patients with wild type KRAS advanced NSCLC
* Determine the clinical response rate (PR (partial response) + CR (complete response)) either monotherapy AZD6244 or the combination AZD6244 plus erlotinib in patients with mutated KRAS advanced NSCLC
* Evaluate disease control rate (PR+CR+SD (stable disease)) and overall survival in both patient groups.
* Determine a safety profile for use of AZD6244 in combination with erlotinib in patients with advanced NSCLC.
* Measure serological markers to evaluate if these markers are correlated with tumor response.
* Measure changes in a tumors MIB-1 (Ki-67) rate and pERK levels in response to treatment with AZD6244.

Eligibility:

* Patients with pathologically confirmed NSCLC not amenable to potentially curative therapy and having progressed after being treated with at least one prior platinum containing chemotherapy regimen, or having refused cytotoxic chemotherapy.
* Progressive disease should be documented prior to enrollment on the study.
* Patient should not have more than 2 prior chemotherapy regimens.
* Measurable disease by RECIST (Response Evaluation Criteria in Solid Tumors) criteria.
* Adequate renal, cardiac, hepatic and hematopoietic functions
* No major surgery, radiotherapy, or chemotherapy within 28 days of enrollment.

Design:

* Patients will be stratified on the basis on their KRAS mutational status. Wild-Type KRAS patients will be randomized to receive either single agent erlotinib 150 mg/day or the combination of erlotinib 100 mg/day plus AZD6244 at 150 mg/day. KRAS mutant patients will be randomized to receive AZD6244 monotherapy at a dose of 75 mg twice per day, or the combination AZD6244 at 150 mg/day plus erlotinib 100 mg/day.
* Treatment will continue until disease progression.
* Toxicity will be assessed every cycle by the CTCAE (Common Terminology Criteria for Adverse Events) Version 4.0.
* Tumor assessments by RECIST 1.1 criteria will be performed every 2 cycles (one cycle is 28 days).
* Correlative studies including initial tumor mutational analysis and tissue immunohistochemistry (IHC) studies will be done on existing tumor blocks, or re-biopsied tissue prior to enrollment.
* Patients will be evaluated for the potential to undergo repeat tumor biopsy after 1 cycle of therapy. Tumors will be assessed for MIB-1 (Ki-67) and pERK levels by IHC.
* The study will accrue up to 40 patients with wild-type KRAS NSCLC and up to 60 patients with mutated KRAS NSCLC.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed advanced (Stage IV) Non Small Cell Lung Cancer that has been verified by the enrolling institution s pathology department. Mixed histologies, with small cell lung cancer components are not eligible.
* Patients must have measurable disease by RECIST criteria, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral CT (computed tomography) scan.
* Patients must have had at least one prior platinum-containing chemotherapy regimen, or have refused cytotoxic chemotherapy. Patients should have no more than two prior chemotherapy regimens. Chemotherapy regimens have no limit on the maximum or minimum number of cycles. Patients enrolled on the trial should have completed their last chemotherapy regimen at least 4 weeks ago. Patients should have completed radiation therapy at least 4 weeks prior to enrollment. Adjuvant and neoadjuvant chemotherapy does not count as prior chemotherapy for advanced disease if more than a year before enrollment.
* Age greater than or equal to 18 years, because no dosing or adverse event data are currently available on the use of AZD6244 (ARRY-142886) as monotherapy or in combination with erlotinib in patients less than 18 years of age. Children are excluded from this study but will be eligible for future pediatric phase 2 combination trials.
* Life expectancy of greater than 3 months.
* ECOG (Eastern Cooperative Oncology Group) performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).
* Patients must have normal organ and marrow function as defined below:

  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin within normal institutional limits
  * AST (aspartate aminotransferase) (SGOT (serum glutamic oxaloacetic transaminase)) /ALT (alanine aminotransferase) ((SGPT (serum glutamic pyruvic transaminase)) less than or equal to 2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits

OR

* creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must have adequate archival material from a previous biopsy to determine KRAS status at the time of enrollment, or undergo a biopsy of fresh tissue of the primary cancer lesion or a metastatic site in order to make this determination.

  * The effects of AZD6244 and erlotinib on the developing human fetus at the recommended therapeutic dose are unknown. However preclinical data showing adverse effects on fetal survival and development with AZD6244 have been reported. For this reason since there is a potential risk of teratogenicity, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and for four weeks after dosing with AZD6244 ceases. Women of child-bearing potential must have a negative pregnancy test prior to entry. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Please note that the AZD6244 manufacturer recommends that adequate contraception for male patients should be used for 16 weeks post-last dose due to sperm life cycle.
  * Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered to less than or equal to grade 1 toxicities from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* In general, patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However, patients who have completed primary treatment of their brain metastasis by surgery or radiotherapy and have been off steroids (with the exception of maintenance replacement steroids) and anti-seizure medications for greater than one month without progression of neurological symptoms are eligible for enrollment in this trial. Stability of treated brain metastases should be confirmed by repeat imaging studies (CT brain or MRI (magnetic resonance imaging) brain) performed at least one month after completion of treatment.
* Previous MEK (methyl ethyl ketone) inhibitor or prior treatment with EGFR TKI (tyrosine kinase inhibitor).
* Major surgery or significant traumatic injury occurring within 21 days prior to treatment.
* Abnormalities of the cornea based on history (e.g., dry eye syndrome, Sjogrens syndrome), congenital abnormality (e.g., Fuchs dystrophy), abnormal slit-lamp examination using a vital dye (e.g., fluorescein, Bengal-Rose), and/or an abnormal corneal sensitivity test (Schirmer test or similar tear production test).
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV (intravenous) alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease.
* Patients with uncontrolled hypertension already on optimal medication, patients with class II or greater heart failure, any current or prior history of cardiomyopathy. Patient with baseline LVEF (left ventricular ejection fraction) less than 50%, atrial fibrillation, recent myocardial infarction, or unstable ischemic heart disease.
* Patients with QTc (corrected QT interval) interval greater than 450 msecs or other factors that increase the risk of QT (Q wave, T wave) prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) including heart failure that meets New York Heart Association (NYHA) class III and IV definitions are excluded. This does not include QTc prolongation secondary to a paced rhythm. If a patient has a paced rhythm, QTc levels less than or equal to 500 (Grade 1) are allowed and patients with QTc > 500 are excluded.
* Required use of a concomitant medication that can prolong the QT interval. A comprehensive list of agents with the potential to cause QTc prolongation can be found at http://www.arizonacert.org/medical-pros/drug-lists/drug-lists.htm.
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g. inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, Hepatitis B or C, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because AZD6244 is a MEK- Inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD6244, breastfeeding should be discontinued if the mother is treated with AZD6244. These potential risks may also apply to other agents used in this study.
* HIV (human immunodeficiency virus) -positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD6244. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

INCLUSION OF WOMEN AND MINORITIES:

Both men and women and members of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-10-26 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2015-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (5):
- United States (5):
  - University of California, Davis, Davis, California
  - University of Southern California Health Sciences Campus, Los Angeles, California
  - City of Hope Medical Group, South Pasadena, California
  - University of Chicago Medical Center, Chicago, Illinois
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ. Cancer statistics, 2009. CA Cancer J Clin. 2009 Jul-Aug;59(4):225-49. doi: 10.3322/caac.20006. Epub 2009 May 27. PMID 19474385
- [Background] Carbone DP, Minna JD. Chemotherapy for non-small cell lung cancer. BMJ. 1995 Oct 7;311(7010):889-90. doi: 10.1136/bmj.311.7010.889. No abstract available. PMID 7580533
- [Background] Rodriguez J, Cortes J, Calvo E, Azinovic I, Fernandez-Hildago O, Martinez-Monge R, Garzon C, de Irala J, Martinez-Aguillo M, Ramon Y Cajal T, Brugarolas A. Paclitaxel, cisplatin, and gemcitabine combination chemotherapy within a multidisciplinary therapeutic approach in metastatic nonsmall cell lung carcinoma. Cancer. 2000 Dec 15;89(12):2622-9. doi: 10.1002/1097-0142(20001215)89:123.0.co;2-x. PMID 11135224
- [Derived] Carter CA, Rajan A, Keen C, Szabo E, Khozin S, Thomas A, Brzezniak C, Guha U, Doyle LA, Steinberg SM, Xi L, Raffeld M, Tomita Y, Lee MJ, Lee S, Trepel JB, Reckamp KL, Koehler S, Gitlitz B, Salgia R, Gandara D, Vokes E, Giaccone G. Selumetinib with and without erlotinib in KRAS mutant and KRAS wild-type advanced nonsmall-cell lung cancer. Ann Oncol. 2016 Apr;27(4):693-9. doi: 10.1093/annonc/mdw008. Epub 2016 Jan 22. PMID 26802155
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-C-0218.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 89 participants were enrolled and 79 participants started. 10 patients should be classified as screen failures. Of the 10, one died during the screening process, and one patient withdrew during the screening process.
Groups:
- KRAS Mut 2: KRAS Mutant patients randomized to combination therapy arm
  AZD6244 + Erlotinib: For KRAS mutant patients and Wild-Type KRAS patients randomized to the combination arm (arms are stratified based on KRAS mutational status), AZD6244 150 mg qd (every day) + erlotinib mg qd.
- WT KRAS 1: Wild-Type KRAS patients randomized to monotherapy arm
  Erlotinib: For Wild-Type KRAS patients randomized to the single agent arm, Erlotinib 150 mg qd
- WT KRAS 2: Wild-Type KRAS patients randomized to combination therapy arm
  AZD6244 + Erlotinib: For KRAS mutant patients and Wild-Type KRAS patients randomized to the combination arm (arms are stratified based on KRAS mutational status), AZD6244 150 mg qd + erl mg qd.
Period: Overall Study
Arm/Group | KRAS Mut 2 | KRAS Mut 1 | WT KRAS 1 | WT KRAS 2
Started | 30 | 11 | 19 | 19
Completed | 28 | 9 | 19 | 19
Not Completed | 2 | 2 | 0 | 0
Not completed — Toxicity | 2 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KRAS Mut 2 | KRAS Mut 1 | WT KRAS 1 | WT KRAS 2 | Total
Number analyzed (Participants) | 30 | 11 | 19 | 19 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 5 | 11 | 10 | 42
  >=65 years | 14 | 6 | 8 | 9 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.05 (9.648) | 64.31 (13.76) | 63.75 (13.6) | 64.84 (8.10) | 65.22 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 7 | 9 | 6 | 38
  Male | 14 | 4 | 10 | 13 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 3 | 8
  Not Hispanic or Latino | 25 | 9 | 15 | 12 | 61
  Unknown or Not Reported | 4 | 0 | 2 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 4 | 4 | 13
  White | 26 | 8 | 14 | 13 | 61
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 11 | 19 | 19 | 79
Histology [Count of Participants; unit: Participants]
  Lung Cancer Adenocarcinoma | 30 | 11 | 15 | 15 | 71
  Squamous cell | 0 | 0 | 4 | 4 | 8
Mutational Status [Count of Participants; unit: Participants] — EGFR (epidermal growth factor receptor); KRAS (Kirsten Rat Sarcoma Viral Oncogene homolog). KRAS G12A (e.g. G is glycine, 12 is the codon or position and A is amino acid alanine); C is cysteine, D is aspartic acid, K is lysine, R is arginine, S is serine, V is valine, Q is glutamine, H is histidine, and L is leucine.
  Participants
    EGFR Mutated (L858R) | 30 | 11 | 1 | 1 | 43
    EGFR Wild Type | 0 | 0 | 18 | 18 | 36
    KRAS G12A | 6 | 0 | 0 | 0 | 6
    KRAS G12C | 8 | 4 | 0 | 0 | 12
    KRAS G12D | 1 | 1 | 0 | 0 | 2
    KRAS G12K | 1 | 1 | 0 | 0 | 2
    KRAS G12R | 0 | 1 | 0 | 0 | 1
    KRAS G12S | 1 | 0 | 0 | 0 | 1
    KRAS G12V | 9 | 4 | 0 | 0 | 13
    KRAS Q61H | 2 | 0 | 0 | 0 | 2
    KRAS Q61L | 2 | 0 | 0 | 0 | 2
    KRAS | 0 | 0 | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — ECOG Performance Status criteria: Grade 0 is normal activity. Fully active, able to carry on all pre-disease performance without restriction. Grade 1 is symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work). Grade 2 is in bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    0 | 3 | 1 | 2 | 2 | 8
    1 | 14 | 5 | 11 | 7 | 37
    2 | 13 | 5 | 6 | 10 | 34
No. of Prior Regimens [Count of Participants; unit: Participants]
  1 | 12 | 6 | 10 | 8 | 36
  2 | 18 | 5 | 9 | 11 | 43
Smoking [Count of Participants; unit: Participants]
  Current | 9 | 0 | 0 | 0 | 9
  Former | 21 | 11 | 13 | 16 | 61
  Never-smoker | 0 | 0 | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Time between the first day of treatment to the day of disease progression. Progressive disease is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that's the smallest on study). In addition to the relative increase of 20% of at least 5mm. (Note: the appearance of one or more lesions is also considered progression).
Time Frame: 2.1 to 4 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | KRAS Mut 2 | KRAS Mut 1 | WT KRAS 1 | WT KRAS 2
Number analyzed (Participants) | 30 | 11 | 19 | 19
Months | 2.3 [2.0 to 4.6] | 4.0 [2.9 to 7.8] | 2.4 [1.3 to 3.7] | 2.1 [1.8 to 5.1]
Statistical Analysis 1: Comparison: KRAS Mut 2 vs KRAS Mut 1; Test type: Superiority or Other; p = 0.24, Log Rank
Statistical Analysis 2: Comparison: WT KRAS 1 vs WT KRAS 2; Test type: Superiority or Other; p = 0.75, Log Rank

2. Primary Outcome: Objective Response
Description: Objective response is complete response + partial response. Complete response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 37 months
Population: There were no partial or complete responses in the KRAS mut 1 arm.
Measure: Number; unit: participants
Arm/Group | KRAS Mut 2 | KRAS Mut 1 | WT KRAS 1 | WT KRAS 2
Number analyzed (Participants) | 30 | 11 | 19 | 19
participants | 3 | 0 | 1 | 2

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 42 months
Population: The combination of toxicities allows for a more robust understanding of the combined therapy toxicities. The dosage of the combination of erlotinib plus AZD6244 was the same whether the pt has a KRAS mutation versus KRAS wild type. KRAS is a molecular mutation and does not change whether or not a pt has toxicities to the combination of therapies.
Measure: Number; unit: Participants
Groups:
- KRAS Mut 2 & WT KRAS 2: KRAS Mutant patients randomized to combination therapy arm
  AZD6244 + Erlotinib: For KRAS mutant patients and Wild-Type KRAS 2 patients randomized to the combination arm (arms are stratified based on KRAS mutational status), AZD6244 150 mg qd (every day) + erlotinib mg qd.
Arm/Group | KRAS Mut 2 & WT KRAS 2 | KRAS Mut 1 | WT KRAS 1
Number analyzed (Participants) | 49 | 11 | 19
Participants | 49 | 9 | 18

4. Secondary Outcome: Percentage of Participants With Disease Control/Stabilization
Description: Disease control/stabilization is the percentage of participants with partial response (PR) + complete response (CR) + stable disease (SD). Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. (Note: the appearance of one or more new lesions is also considered progressions.), taking as reference the smallest sum diameters.
Time Frame: 3 cycles or up to 84 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | KRAS Mut 2 | KRAS Mut 1 | WT KRAS 1 | WT KRAS 2
Number analyzed (Participants) | 30 | 11 | 19 | 19
percentage of participants | 43 [25.5 to 52.6] | 89 [51.8 to 99.7] | 47 [24.4 to 71.1] | 35.3 [14.2 to 61.7]

5. Secondary Outcome: Overall Survival
Description: Time between the first day of treatment to the time of death.
Time Frame: Up to 26 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | KRAS Mut 2 | KRAS Mut 1 | WT KRAS 1 | WT KRAS 2
Number analyzed (Participants) | 30 | 11 | 19 | 19
Months | 21.8 [5.7 to NA] — The upper end of the confidence interval is undefined because there were too few events to calculate. | 10.5 [5.7 to NA] — The upper end of the confidence interval is undefined because there were too few events to calculate. | 6.3 [2.6 to 19.5] | 12.9 [3.5 to 25.4]
Statistical Analysis 1: Comparison: WT KRAS 1 vs WT KRAS 2; Test type: Superiority or Other; p = 0.51, Log Rank
Statistical Analysis 2: Comparison: KRAS Mut 2 vs KRAS Mut 1; Test type: Superiority or Other; p = 0.81, Log Rank

6. Secondary Outcome: Percentage of Th17 in Cluster of Differentiation 4 (CD4)+T Cells at Baseline in Relation to Response
Description: First the number of T cells that are CD4+ is determined by staining with an antibody to CD4 and measured in a flow cytometer. Then the number of Th17+ cells is determined by staining with an antibody to IL-17 and measured in a flow cytometer. Then the percentage of CD4+ cells that are also Th17 cells is determined as a simple ratio, i.e. Th17cells/CD4 cells. This ratio is reported here for each category of KRAS mutation status for whom we had patients.
Time Frame: Pretreatment - Cycle 1 Day 1
Population: No participants were analyzed in the WT KRAS 1 cohort because no samples were available for analysis. For all other cohorts, the numbers analyzed indicates some samples were either not drawn or could not be located.
Measure: Mean (Standard Deviation); unit: Percentage of Th17 in CD4+T Cells
Arm/Group | KRAS Mut 2 | KRAS Mut 1 | WT KRAS 2
Number analyzed (Participants) | 15 | 4 | 9
Percentage of Th17 in CD4+T Cells | 0.19 (0.18) | 0.11 (0.05) | 0.34 (0.27)

7. Secondary Outcome: Number of Participants With a Reduction in Phosphorylated Extracellular Signal-Regulated Kinases (p-ERK) in Lymphocytes
Description: Level of p-ERK was measured by the median channel cumber of fluorescence intensity. Data are relative to the level before therapy begins(C1D1).Then we see what the level was after therapy & compare. Every value after therapy is compared to pre-therapy, & every patient is their own control. To do that, we make C1D1 equal to 1 for every patient & then compare the pERK level after therapy by looking at the fold change in pERK level.
Time Frame: Cycle 1 Day 1 pre-treatment with Cycle 1 Day 2 (1 day after starting treatment), and Cycle 1 Day 14 (2 weeks after starting treatment)
Population: Re: number of participants analyzed: Samples were either not drawn or could not be located. WT KRAS 1/WT KRAS 2 are missing because the effect of treatment on the Ras-Raf-MEK-ERK pathway as measured by a reduction in phosphorylated extracellular signal-regulated kinases (p-ERK) in lymphocytes was evaluated in patients with KRAS-mutated tumors only.
Measure: Number; unit: participants
Arm/Group | KRAS Mut 2 | KRAS Mut 1
Number analyzed (Participants) | 17 | 4
participants
  Cycle 1 Day 1 | NA — C1D1 is NA because every other time point, pERK level was normalized against C1D1; all the C1D1 values were set to 1. | NA — C1D1 is NA because every other time point, pERK level was normalized against C1D1; all the C1D1 values were set to 1.
  Cycle 1 day 2 | 17 | 4
  Cycle 1 day 14 | 14 | 2
Statistical Analysis 1: Comparison: KRAS Mut 1; Test type: Superiority or Other; p < 0.0007, Wilcoxon matched-pairs signed rank test — P-value was determined by comparison by the level of p-ERK at cycle 1 day 1 to cycle 1 day 2
Statistical Analysis 2: Comparison: KRAS Mut 1; Test type: Superiority or Other; p < 0.0001, Wilcoxon matched-pairs signed rank test — P-value was determined by comparison by the level of p-ERK at cycle 1 day 1 to cycle 1 day 14
Statistical Analysis 3: Comparison: KRAS Mut 1; 4 patients in this group; statistically underpowered; Test type: Superiority or Other; p = 0.0209, Wilcoxon matched-pairs signed rank test — P-value was determined by comparison by the level of p-ERK at cycle 1 day 2 and cycle 1 day 14

8. Other Pre Specified Outcome: Number of Participants With Changes in a Tumor's MIB-1 (Ki-67) Rate
Description: Changes in a tumor's MIB-1 (Ki-67) rate was to be assessed by immunohistochemistry.
Time Frame: At enrollment
Population: Tumor MIB-1 (Ki-67) rate testing was not done because it was too costly.
Arm/Group | KRAS Mut 2 | KRAS Mut 1 | WT KRAS 1 | WT KRAS 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Other Pre Specified Outcome: Change in T Cell Immunoglobulin Mucin 3 (TIM-3) on Tregs
Description: Fold change from cycle 1 day 1 was determined by TIM-3 expression level on Tregs measured by the median channel number of fluorescence intensity.
Time Frame: as for outcome 7
Population: These are exploratory results and a normal range has not been defined for fold change. No participants were analyzed in the WT KRAS 1 cohort because no samples were available for analysis. Missing numbers in the other cohorts were either not drawn, misplaced or the samples were not viable.
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | KRAS Mut 2 | KRAS Mut 1 | WT KRAS 2
Number analyzed (Participants) | 17 | 4 | 8
Fold change
  Cycle 1 Day 2 | 1.01 (0.09) | 1.01 (0.12) | 1.11 (0.13)
  Cycle 1 Day 14 | 0.98 (0.10) | 0.84 (0.07) | 0.96 (0.11)

10. Other Pre Specified Outcome: Change in Cytotoxic T-lymphocyte Associated Protein 4 (CTLA-4) Expression on Tregs
Description: The fold change from cycle 1 day 1 was determined by the level of CTLA-4 expression on Tregs measured by the median channel number of fluorescence intensity.
Time Frame: as for outcome 7
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | KRAS Mut 2 | KRAS Mut 1 | WT KRAS 2
Number analyzed (Participants) | 17 | 4 | 10
Fold change
  Cycle 1 Day 2 | 0.95 (0.17) | 0.85 (0.10) | 1.15 (0.28)
  Cycle 1 Day 14 | 1.25 (0.46) | 0.89 (0.29) | 1.49 (0.61)

11. Other Pre Specified Outcome: Change in Programmed Cell Death-1 (PD-1) Expression on Tregs
Description: Fold change from cycle 1 day 1 was determined by the PD-1 expression level on Tregs measured by the median channel number of fluorescence intensity.
Time Frame: as for outcome 7
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | KRAS Mut 2 | KRAS Mut 1 | WT KRAS 2
Number analyzed (Participants) | 17 | 4 | 10
Fold change
  Cycle 1 Day 2 | 0.99 (0.28) | 0.96 (0.09) | 1.33 (0.57)
  Cycle 1 Day 14 | 1.31 (0.42) | 0.98 (0.04) | 2.31 (1.77)

12. Other Pre Specified Outcome: Change in Programmed Cell Death-1 (PD-1) Expression on Cluster of Differentiation 8 (CD8)+T Cells
Description: Fold change from cycle 1 day 1 was determined by programmed cell death-1 (PD-1) expression on CD8+ T cells measured by the median channel number of fluorescence intensity.
Time Frame: as for outcome 7
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | KRAS Mut 2 | KRAS Mut 1 | WT KRAS 2
Number analyzed (Participants) | 17 | 4 | 10
Fold change
  Cycel 1 Day 2 | 1.05 (0.15) | 1.09 (0.33) | 1.19 (0.40)
  Cycle 1 Day 14 | 1.16 (0.27) | 1.14 (0.34) | 1.26 (0.25)

13. Other Pre Specified Outcome: Phospho-ERK (p-ERK), Phospho Protein Kinase B (p-AKt) and Phosphatase and Tensin Homolog (PTEN) Expression Testing
Description: p-ERK, p-AKt and PTEN protein expression testing was to be assessed by immunohistochemistry.
Time Frame: At enrollment
Population: Zero participants were analyzed because most of the immunohistochemistry (IHC) specialty assays (e.g. IHC, fluoresense in situ hybridization (FISH), polymerase chain reaction (PCR) were not available (still are not performed in path) and required funding for development that was not provided.
Arm/Group | KRAS Mut 2 | KRAS Mut 1 | WT KRAS 1 | WT KRAS 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Other Pre Specified Outcome: Number of Participants With Overexpression of Estimated Glomerular Filtration Rate (EGFR) and c-MET
Description: Number of participants with over expression of EGFR and c-MET was to be assessed by fluoresense in situ hybridization (FISH).
Time Frame: At enrollment
Population: as for outcome 13
Arm/Group | KRAS Mut 2 | KRAS Mut 1 | WT KRAS 1 | WT KRAS 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Other Pre Specified Outcome: Number of Participants Who Underwent Mutational Analysis for Estimated Glomerular Filtration Rate (EGFR), Mitogen-activated Protein Kinase 1 (MEK 1), Proto-oncogene B-Raf (BRAF), and LKB1
Description: Number of participants who underwent mutational analysis for EGFR, MEK 1, BRAF, and LKB1 was to be assessed by polymerase chain reaction (PCR).
Time Frame: At enrollment
Population: as for outcome 13
Arm/Group | KRAS Mut 2 | KRAS Mut 1 | WT KRAS 1 | WT KRAS 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The combination of toxicities allows for a more robust understanding of the combined therapy toxicities. The dosage of the combination of erlotinib plus AZD6244 was the same whether the pt has a KRAS mutation versus KRAS wild type. KRAS is a molecular mutation and does not change whether or not a pt has toxicities to the combination of therapies.
Arm/Group | KRAS Mut 2 & WT KRAS 2 | KRAS Mut 1 | WT KRAS 1
All-Cause Mortality (participants affected / at risk) | 17/49 | 4/11 | 8/19
Serious Adverse Events (participants affected / at risk) | 30/49 | 6/11 | 11/19
Other Adverse Events (participants affected / at risk) | 49/49 | 9/11 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KRAS Mut 2 & WT KRAS 2 (N=49) | KRAS Mut 1 (N=11) | WT KRAS 1 (N=19)
Death NOS (General disorders) | 16 (16) | 4 (4) | 8 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 2 (2)
INR increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (6) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (left ventricular systolic dysfunction) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — sudden left leg numbness
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 2 (2) — (inclu cysts and polyps) - Other specify (death)
Gastrointestinal disorders - Other, specify (bile duct obstruction) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 0 (0) — progressive disease; disease progression
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KRAS Mut 2 & WT KRAS 2 (N=49) | KRAS Mut 1 (N=11) | WT KRAS 1 (N=19)
Abdominal pain (Gastrointestinal disorders) | 9 (11) | 1 (2) | 3 (4)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3) | 1 (1) | 2 (4)
Alanine aminotransferase increased (Investigations) | 27 (51) | 5 (7) | 4 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 24 (54) | 4 (4) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 17 (23) | 4 (4) | 9 (10)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 34 (65) | 5 (10) | 4 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 13 (16) | 0 (0) | 2 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
CPK increased (Investigations) | 15 (39) | 5 (10) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 4 (4) | 1 (2) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 1 (1)
Chills (General disorders) | 7 (8) | 0 (0) | 3 (3)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 6 (7) | 5 (9) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 2 (2) | 9 (16)
Creatinine increased (Investigations) | 13 (19) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 43 (94) | 4 (6) | 8 (16)
Dry eye (Eye disorders) | 6 (7) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 6 (7) | 3 (3) | 3 (3)
Dysgeusia (Nervous system disorders) | 12 (13) | 1 (1) | 1 (3)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 7 (9) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 4 (7) | 7 (8)
Edema limbs (General disorders) | 19 (26) | 6 (10) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Fatigue (General disorders) | 25 (47) | 2 (4) | 6 (7)
Fever (General disorders) | 6 (6) | 1 (1) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Floaters (Eye disorders) | 2 (3) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (4) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 9 (12) | 0 (0) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (3)
Hypertension (Vascular disorders) | 8 (15) | 0 (0) | 2 (4)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 36 (64) | 7 (9) | 5 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 5 (6) | 0 (0) | 2 (7)
Hypokalemia (Metabolism and nutrition disorders) | 11 (13) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 19 (29) | 3 (5) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 22 (31) | 0 (0) | 4 (11)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (15) | 1 (2) | 4 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 2 (2)
Infections and infestations-Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — urinary tract infection
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1) | 2 (2)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 21 (56) | 1 (1) | 8 (9)
Mucositis oral (Gastrointestinal disorders) | 11 (15) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 27 (48) | 3 (5) | 9 (11)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Other, specify (progressive disease)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0) | 2 (2)
Pain (General disorders) | 10 (12) | 3 (4) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Paresthesia (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 9 (13) | 0 (0) | 2 (4)
Platelet count decreased (Investigations) | 14 (23) | 3 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 12 (14) | 1 (1) | 5 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 22 (39) | 4 (5) | 8 (14)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 27 (51) | 4 (6) | 8 (12)
Renal and urinary disorders - Other, specify (urinary burning) (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Runny nose, non allergy
Sinus tachycardia (Cardiac disorders) | 7 (7) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders-Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (6) — dermatitis, rash in peri-anal area; erythematous rash; ingrown toenail; L arm abrasions from fall; nail overgrowth; erythema on the nose
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 6 (6) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 0 (0) | 2 (3)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 19 (38) | 1 (1) | 2 (2)
Weight loss (Investigations) | 10 (12) | 0 (0) | 2 (2)
Alkaline phosphatase increased (Investigations) | 13 (19) | 3 (4) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) — diastolic dysfunction
Edema face (General disorders) | 4 (6) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 6 (7) | 2 (4) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6) | 2 (3) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2) | 1 (3) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — left foot numbness
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 8 (9) | 2 (5) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Other, specify (decreased breath sounds)
Dry skin (Skin and subcutaneous tissue disorders) | 19 (21) | 2 (2) | 6 (9)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 10 (13) | 0 (0) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 6 (8) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 13 (14) | 0 (0) | 0 (0)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders- Other, specify (Eye disorders) | 4 (5) | 0 (0) | 0 (0) — decreased vision; eye lash thickening; glare; left lower eyelid excoriation; red, green eyes spots
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 2 (2) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 2 (3) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (bloody stools) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
General disorders and adminstration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0) — Feverish
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (6) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (4) | 0 (0) | 0 (0)
Hypothryoidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — intolerance to cold
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — sensitivity to cold
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0 (0)
Periorbital infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (emotional) (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — diminished breath sounds
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) — contact dermatitis; skin eczematous dry patches on dorsum of both feet; skin bleeding
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No